CLINICAL TRIAL: NCT04467840
Title: Opaganib, a Sphingosine Kinase-2 (SK2) Inhibitor in COVID-19 Pneumonia: a Randomized, Double-blind, Placebo-Controlled Phase 2/3 Study, in Adult Subjects Hospitalized With Severe SARS-CoV-2 Positive Pneumonia
Brief Title: Opaganib, a Sphingosine Kinase-2 (SK2) Inhibitor in COVID-19 Pneumonia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: RedHill Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABC-201
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Results first posted 2023-10-19 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: COVID-19; Lung Infection
Keywords: Therapeutic Use
MeSH Terms: conditions — COVID-19 | interventions — 3-(4-chlorophenyl)-adamantane-1-carboxylic acid (pyridin-4-ylmethyl)amide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Opaganib (Experimental): In addition to standard of care, opaganib will be administered orally with 2 x 250 mg capsules (500 mg) every 12 hours. When required this may be made into a suspension form and may be administered by nasogastric tube.
  Interventions: Drug: Opaganib
- Placebo (Placebo Comparator): In addition to standard of care, a matching placebo will be administered orally with 2 x 250 mg capsules (500 mg) every 12 hours. Where required this may be made into a suspension form and may be administered by nasogastric tube.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Opaganib — Study participants will receive either opaganib 2 x 250 mg capsules (500 mg) every 12 hours, or matching placebo, in addition to standard of care (pharmacological as defined above and/or supportive) at any given institution. Study drug will be administered every day for 14 days (Day 1 to Day 14).
  Other Names: Yeliva; ABC294640
  Arms: Opaganib
Drug: Placebo — Study participants will receive either opaganib 2 x 250 mg capsules (500 mg) every 12 hours, or matching placebo, in addition to standard of care (pharmacological as defined above and/or supportive) at any given institution. Study drug will be administered every day for 14 days (Day 1 to Day 14).
  Arms: Placebo

SUMMARY:
A phase 2/3 multi-center randomized, double-blind, parallel arm, placebo- controlled study in Adult Subjects Hospitalized with Severe SARS-CoV-2 Positive Pneumonia to determine the potential of opaganib to improve and/or stabilize the clinical status of the patient.

DETAILED DESCRIPTION:
This is a phase 2/3 multi-center randomized, double-blind, parallel arm, placebo- controlled study with an adaptive design that will utilize a futility assessment. The study is planned be performed worldwide in up to approximately 80 clinical sites.

After informed consent is obtained, patients will enter a screening phase for no more than 3 days, to determine eligibility. Approximately 464 eligible patients will be randomized and receive either opaganib added to standard of care, or matching placebo added to standard of care, in a randomization ratio of 1:1. Treatment assignments will remain blinded to the patient, investigator and hospital staff, as well as the sponsor. As the approval and/or guidance for treating COVID-19 are evolving, for this protocol, standard of care will be defined by the recommended schemes of treatment according to the severity of the disease, taking into consideration regulatory approvals in one or more regions.

Study participants will receive either opaganib 2 x 250 mg capsules (500 mg) every 12 hours, or matching placebo, in addition to standard of care (pharmacological as defined above and/or supportive) at any given institution. Study drug will be administered every day for 14 days (Day 1 to Day 14). All participants will be followed up for 28 days after their last dose of study drug, which may occur at Day 14 or after premature study drug discontinuation, based upon patient or physician determination.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female ≥18 to ≤80 years of age
2. Proven COVID-19 infection per RT-PCR assay of a pharyngeal sample (nasopharyngeal or oropharyngeal) AND pneumonia defined as radiographic opacities on chest X-ray or CT scan. that diagnosed COVID-19 pneumonia. Pharyngeal samples collected either at screening or within 7-days prior to screening for the same ongoing COVID-19 pneumonia illness are acceptable
3. The patient requires, at baseline, high flow supplemental oxygen or positive pressure ventilation or is receiving oxygen via face mask, such as a non-rebreather or reservoir mask, capable of delivering high concentrations of oxygen
4. Patient agrees to use appropriate methods of contraception during the study and 3 months after the last dose of study drug
5. The patient or legal representative has signed a written informed consent approved by the IRB/Ethics Committee

Exclusion Criteria:

1. Any co-morbidity that may add risk to the treatment in the judgment of the investigator, particularly patients with known cardiac conditions, and serious neuropsychiatric conditions such as psychosis or major depression
2. Requiring intubation and mechanical ventilation at baseline
3. Patient has a 'Do Not Intubate' and/or 'Do Not Resuscitate' order in place
4. Oxygen saturation >95% on room air
5. Any preexisting respiratory condition that requires intermittent or continuous ambulatory oxygen prior to hospitalization
6. Patient is, in the investigator's clinical judgement, unlikely to survive >72 hours
7. Pregnant (positive serum or urine test within 3 days prior to randomization) or nursing women .
8. Unwillingness or inability to comply with procedures required in this protocol.
9. Corrected QT (QTc) interval on electrocardiogram (ECG) >470 ms for females or >450 ms for males, calculated using Friedericia's formula (QTcF)
10. AST (SGOT) or ALT (SGPT) > 2.0 x upper limit of normal (ULN)
11. Total bilirubin >1.5x ULN (except where bilirubin increase is due to Gilbert's Syndrome)
12. Serum creatinine >2.0 X ULN
13. Absolute neutrophil count <1000 cells/mm3
14. Platelet count <75,000/mm3
15. Hemoglobin <8.0 g/dL
16. Medications that are sensitive substrates, or substrates with a narrow therapeutic range, for CYP1A2, CYP2B6, CYP2C8, CYP2C9, CYP2C19 CYP2D6 , CYP3A4, P-gP, BCRP and OATP1B1 should be avoided with opaganib
17. Moderate or strong inhibitors of CYP1A2, CYP3A4, CYP2D6 or P-gP or moderate to strong inducers of CYP3A4 and CYP1A2 are prohibited
18. Currently taking warfarin, apixaban, argatroban or rivaroxaban due to drug-drug interaction based on CYP450 metabolism
19. Current drug or alcohol abuse
20. Currently participating in a clinical study assessing pharmacological treatments, including anti-viral studies
21. Treatment with any medication that causes QT prolongation within seven days, or 5 half-lives, whichever is longest, prior to initiation of study drug, or intention to use them throughout the study, including but not limited to: amiodarone, amitriptyline, citalopram dose greater than 20 mg/day, dihydroergotamine, disopyramide, dofetilide, dronedarone, ergotamine, ibutilde, ondansetron or other 5-HT3 receptor antagonists, pimozide, procainamide, quinidine, quinine, quinolone, ranolazine, risperidone, sotaloland tolteridine. Investigators are directed to the following up-to-date web site listing QT prolonging drugs: https://www.crediblemeds.org/index.php/drugsearch

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2021-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Levitt, MD, Study Director — RedHill Biopharma Limited
Locations (57):
- ABC-201 Site 901, Detroit, Michigan, United States
- Brazil (10):
  - ABC-201 Site 408, Belo Horizonte
  - ABC-201 Site 411, Belo Horizonte
  - ABC-201 Site 405, Joinville
  - ABC-201 Site 404, Paraná
  - ABC-201 Site 410, Passo Fundo
  - ABC-201 Site 409, Porto Alegre
  - ABC-201 Site 402, São Bernardo do Campo
  - ABC-201 Site 401, São Paulo
  - ABC-201 Site 403, São Paulo
  - ABC-201 Site 407, Tubarão
- Colombia (5):
  - ABC-201 Site 604, Medellín, Antioquia
  - ABC-201 Site 603, Bogotá
  - ABC-201 Site 605, Cundinamarca
  - ABC-201 Site 602, Medellín
  - ABC-201 Site 601, Santiago de Cali
- Israel (8):
  - ABC-201 Site 708, Ashkelon, Ashketon
  - ABC-201 Site 702, Ashdod
  - ABC-201 Site 704, Holon
  - ABC-201 Site 701, Jerusalem
  - ABC-201,Site 709, Kfar Saba
  - ABC-201 Site 705, Nahariya
  - ABC-201 Site 706, Nazareth
  - ABC-201 Site 703, Safed
- Italy (4):
  - ABC-201 Site 203, Alessandria
  - ABC-201 Site 201, Lecco
  - ABC-201 Site 202, Milan
  - ABC-201 Site 204, Torino
- Mexico (2):
  - ABC-201 Site 501, Mexico City
  - ABC-201 Site 503, Sinaloa
- ABC-201 Site 655, Lima, Peru
- Poland (8):
  - ABC-201 Site 303, Bolesławiec
  - ABC-201 Site 306, Katowice
  - ABC-201 Site 304, Koszalin
  - ABC-201 Site 308, Lodz
  - ABC-201 Site 307, Lublin
  - ABC-201 Site 302, Ostróda
  - ABC-201 Site 301, Racibórz
  - ABC-201 Site 305, Wroclaw
- Russia (15):
  - ABC-201 Site 110, Barnaul
  - ABC-201 Site 122, Kirovsk
  - ABC-201 Site 101, Moscow
  - ABC-201 Site 132, Moscow
  - ABC-201 Site 120, Murmansk
  - ABC-201 Site 103, Ryazan
  - ABC-201 Site 114, Ryazan
  - ABC-201 Site 109, Saint Petersburg
  - ABC-201 Site 111, Saint Petersburg
  - ABC-201 Site 129, Saint Petersburg
  - ABC-201 Site 108, Saratov
  - ABC-201 Site 102, Smolensk
  - ABC-201 Site 104, Tver'
  - ABC-201 Site 118, Volgograd
  - ABC-201 Site 112, Yaroslavl
- United Kingdom (3):
  - ABC-201 Site 253, Antrim
  - ABC-201 Site 251, Gillingham
  - ABC-201 Site 252, Taunton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Opaganib | Placebo
Started (ITT populaion) | 237 | 238
mITT Population | 230 | 233
Completed | 186 | 186
Not Completed | 51 | 52
Not completed — Death | 35 | 39
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Other | 1 | 5
Not completed — Missing study completion status | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Opaganib: Opaganib administered orally in 2 x 250 mg capsules (500 mg) every 12 hours every day for 14 days (Day 1 to Day 14) in addition to standard of care. When required this may be made into a suspension form and may be administered by nasogastric tube.
- Placebo: Matching placebo administered orally in 2 x 250 mg capsules (500 mg) every 12 hours every day for 14 days (Day 1 to Day 14) in addition to standard of care. Where required this may be made into a suspension form and may be administered by nasogastric tube.
- Total: Total of all reporting groups
Arm/Group | Opaganib | Placebo | Total
Number analyzed (Participants) | 237 | 238 | 475
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 189 | 169 | 358
  >=65 years | 48 | 69 | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (12.05) | 57.3 (12.74) | 56.5 (12.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 76 | 162
  Male | 151 | 162 | 313
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 9
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 197 | 203 | 400
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 23 | 18 | 41
Region of Enrollment [Number; unit: participants]
  Colombia | 10 | 8 | 18
  Brazil | 61 | 62 | 123
  Poland | 12 | 16 | 28
  Italy | 25 | 28 | 53
  Mexico | 7 | 4 | 11
  Israel | 43 | 40 | 83
  Russia | 79 | 80 | 159
HbA1c at Screening [Count of Participants; unit: Participants]
  <6.5 and not on active treatment with insulin or oral hypoglycemics | 154 | 157 | 311
  ≥6.5 or on active treatment with insulin or oral hypoglycemics | 83 | 80 | 163
  Missing | 0 | 1 | 1
BMI at Baseline (kg/m^2) [Mean (Standard Deviation); unit: kg/m2] — Population: Information reported according to data collected. Where the number of participants analyzed differs from the overall, the data was not collected/reported by the clinical site.
  kg/m2
    number analyzed (Participants) | 223 | 228 | 451
    (all) | 31.02 (5.676) | 30.47 (5.158) | 30.74 (5.421)
Supplemental Oxygen at Baseline [Count of Participants; unit: Participants]
  Yes | 229 | 233 | 462
  No | 1 | 0 | 1
  Missing | 7 | 5 | 12
Oxygen type (for supplemental oxygen at baseline - Yes) [Count of Participants; unit: Participants] — There were 475 participants in the Intent to Treat (ITT) population, but the primary analysis was based on the modified ITT (mITT) population comprised of all participants who received at least one dose of investigational product (IP): n=463. Of these 463 participants, data was missing on 1. Population: Number of subjects on supplemental oxygen at baseline
  Participants
    number analyzed (Participants) | 229 | 233 | 462
    Intubation/Mechanical ventilation | 1 | 2 | 3
    Low Flow Nasal Cannulas (LFNC) | 3 | 1 | 4
    Non-invasive ventilation/High Flow Nasal Cannulas (HFNC)/Mask with reservoir/Mask without reservoir | 225 | 230 | 455
Oxygen flow at baseline (L/min) [Mean (Standard Deviation); unit: L/min] — Population: Baseline oxygen flow was only collected in subjects not intubated at baseline who required oxygen and who had baseline oxygen recorded.
  L/min
    number analyzed (Participants) | 222 | 219 | 441
    (all) | 24.6 (19.59) | 24.9 (19.83) | 24.8 (19.69)
Oxygen in the gas mix (%) [Mean (Standard Deviation); unit: Percentage of oxygen] — Population: Missing data was not collected by the clinical sites
  Percentage of oxygen
    number analyzed (Participants) | 222 | 222 | 444
    (all) | 65.5 (60.0) | 64.1 (60.0) | 64.8 (60.0)
Median percentage of oxygen in the gas mix (%) [Median (Full Range); unit: Percentage of oxygen] — Population: Missing data was not collected by the clinical sites
  Percentage of oxygen
    number analyzed (Participants) | 222 | 222 | 444
    (all) | 60.0 [25 to 100] | 60.0 [30 to 100] | 60.0 [25 to 100]
FiO2≤60% sub-population inflammation markers: lymphocyte counts [Median (Inter-Quartile Range); unit: 10^9*cell/L] — Median baseline levels lymphocyte counts in the "lower FiO2" (FiO2 at baseline ≤ the median of 60%) FiO2 sub-population are presented here Population: A post hoc analysis set comprised two sub-populations, namely, "lower FiO2" (FiO2 at baseline ≤ the median of 60%) and "higher FiO2" (FiO2 at baseline > the median of 60%) was added after the final version of the SAP was signed.
  Missing data was not collected by the clinical sites
  10^9*cell/L
    number analyzed (Participants) | 116 | 133 | 249
    (all) | 0.910 [0.69 to 1.36] | 1.010 [0.72 to 1.41] | 0.990 [0.71 to 1.38]
FiO2≤60% sub-population inflammation markers: CRP Levels [Median (Inter-Quartile Range); unit: mg/L] — FiO2≤60% sub-population inflammation markers:CRP Levels[1][2] Population: Measure Analysis Population Description: A post hoc analysis set comprised two sub-populations, namely, "lower FiO2" (FiO2 at baseline ≤ the median of 60%) and "higher FiO2" (FiO2 at baseline > the median of 60%) was added after the final version of the SAP was signed.
  Missing data was not collected by the clinical sites
  mg/L
    number analyzed (Participants) | 113 | 127 | 240
    (all) | 67.100 [26.77 to 173.00] | 45.00 [18.60 to 145.60] | 60.80 [21.40 to 153.40]
FiO2≤60% sub-population inflammation markers: Ferritin Levels [Median (Inter-Quartile Range); unit: ug/L] — Measure Description: FiO2≤60% sub-population inflammation markers:Ferritin Levels[1][2] Population: Measure Analysis Population Description: Measure Analysis Population Description: A post hoc analysis set comprised two sub-populations, namely, "lower FiO2" (FiO2 at baseline ≤ the median of 60%) and "higher FiO2" (FiO2 at baseline > the median of 60%) was added after the final version of the SAP was signed.
  Missing data was not collected by the clinical sites
  ug/L
    number analyzed (Participants) | 104 | 124 | 228
    (all) | 727.600 [381.65 to 1383.45] | 592.300 [368.02 to 1201.20] | 666.950 [370.17 to 1297.50]
FiO2≤60% sub-population inflammation markers: D-Dimer Levels [Median (Inter-Quartile Range); unit: ug/ml] — Median baseline levels of systemic markers of inflammation -D-Dimer FiO2≤60% sub-population Population: A post hoc analysis set comprised two sub-populations, namely, "lower FiO2" (FiO2 at baseline ≤ the median of 60%) and "higher FiO2" (FiO2 at baseline > the median of 60%) was added after the final version of the SAP was signed
  Missing data was not collected by the clinical sites
  ug/ml
    number analyzed (Participants) | 111 | 129 | 240
    (all) | 0.499 [0.17 to 1.17] | 0.380 [0.18 to 1.04] | 0.450 [0.18 to 1.06]
FiO2≤60% sub-population inflammation markers: Lactate Dehydrogenase [Median (Inter-Quartile Range); unit: IU/L] — Median baseline levels Lactate Dehydrogenase in the "lower FiO2" (FiO2 at baseline ≤ the median of 60%) FiO2 sub-population are presented here Population: A post hoc analysis set comprised two sub-populations, namely, "lower FiO2" (FiO2 at baseline ≤ the median of 60%) and "higher FiO2" (FiO2 at baseline > the median of 60%) was added after the final version of the SAP was signed.
  Missing data was not collected by the clinical sites
  IU/L
    number analyzed (Participants) | 106 | 124 | 230
    (all) | 359.400 [300.00 to 507.00] | 368.750 [287.55 to 536.34] | 361.150 [290.60 to 522.00]
FiO2>60% sub-population lymphocyte counts [Median (Inter-Quartile Range); unit: 10^9*cell/L] — Median baseline levels lymphocyte counts in the "higher FiO2" (FiO2 at baseline > the median of 60%) FiO2 sub-population are presented here Population: Measure Analysis Population Description: A post hoc analysis set comprised two sub-populations, namely, "lower FiO2" (FiO2 at baseline ≤ the median of 60%) and "higher FiO2" (FiO2 at baseline > the median of 60%) was added after the final version of the SAP was signed.
  10^9*cell/L
    number analyzed (Participants) | 105 | 84 | 189
    (all) | 0.840 [0.55 to 1.27] | 0.700 [0.49 to 1.07] | 0.792 [0.50 to 1.20]
FiO2>60% sub-population inflammation markers: CRP levels [Median (Inter-Quartile Range); unit: mg/L] — Median baseline levels CRP levels in the "higher FiO2" (FiO2 at baseline > the median of 60%) FiO2 sub-population are presented here Population: A post hoc analysis set comprised two sub-populations, namely, "lower FiO2" (FiO2 at baseline ≤ the median of 60%) and "higher FiO2" (FiO2 at baseline > the median of 60%) was added after the final version of the SAP was signed.
  Missing data was not collected by the clinical sites
  mg/L
    number analyzed (Participants) | 100 | 86 | 186
    (all) | 94.050 [45.20 to 193.65] | 106.370 [36.50 to 208.84] | 102.800 [38.67 to 200.30]
FiO2>60% sub-population inflammation markers: Ferritin Levels [Median (Inter-Quartile Range); unit: ug/L] — Median baseline levels ferritin levels in the "higher FiO2" (FiO2 at baseline > the median of 60%) FiO2 sub-population are presented here Population: A post hoc analysis set comprised two sub-populations, namely, "lower FiO2" (FiO2 at baseline ≤ the median of 60%) and "higher FiO2" (FiO2 at baseline > the median of 60%) was added after the final version of the SAP was signed.
  Missing data was not collected by the clinical sites
  ug/L
    number analyzed (Participants) | 88 | 79 | 167
    (all) | 1074.150 [590.50 to 1587.12] | 980.00 [445.00 to 2000.00] | 1000.00 [500.60 to 2000.00]
FiO2>60% sub-population inflammation markers: D-Dimer Levels [Median (Inter-Quartile Range); unit: ug/ml] — Median baseline levels D-Dimer levels in the "higher FiO2" (FiO2 at baseline > the median of 60%) FiO2 sub-population are presented here Population: A post hoc analysis set comprised two sub-populations, namely, "lower FiO2" (FiO2 at baseline ≤ the median of 60%) and "higher FiO2" (FiO2 at baseline > the median of 60%) was added after the final version of the SAP was signed.
  Missing data was not collected by the clinical sites
  ug/ml
    number analyzed (Participants) | 94 | 84 | 178
    (all) | 0.790 [0.29 to 1.95] | 0.836 [0.32 to 662.00] | 0.806 [0.31 to 1.79]
FiO2>60% sub-population inflammation markers: Lactate Dehydrogenase Levels [Median (Inter-Quartile Range); unit: IU/L] — Median baseline: Lactate Dehydrogenase levels in the "higher FiO2" (FiO2 at baseline > the median of 60%) FiO2 sub-population are presented here Population: A post hoc analysis set comprised two sub-populations, namely, "lower FiO2" (FiO2 at baseline ≤ the median of 60%) and "higher FiO2" (FiO2 at baseline > the median of 60%) was added after the final version of the SAP was signed.
  Missing data was not collected by the clinical sites
  IU/L
    number analyzed (Participants) | 100 | 83 | 183
    (all) | 477.500 [366.50 to 641.50] | 447.00 [339.00 to 662.00] | 469.230 [344.00 to 644.00]

OUTCOME MEASURES:

1. Primary Outcome: Supplemental Oxygen Requirement
Description: To compare the proportion of patients no longer requiring supplemental oxygen for at least 24 hours by Day 14 between subjects taking opaganib and those on placebo.
Time Frame: 14 days maintained up to 42 days
Population: Modified ITT (mITT) population defined as randomized subjects who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 230 | 233
Participants
  Subjects not receiving supplemental oxygen for at least 24 hours by Day 14 and maintained at Day 42 | 139 | 132
  Subjects receiving supplemental oxygen (including: death, lost to follow-up, or need of oxygen) | 91 | 101
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.391, Cochran-Mantel-Haenszel — The threshold for statistical significance was p = 0.05; Risk Difference (RD) = 3.86, 95% CI 2-sided [-4.93 to 12.65] — Opaganib - Placebo

2. Secondary Outcome: Percentage of Subjects With ≥ 2 Category Improvement on the World Health Organization (WHO) Ordinal Scale for Clinical Improvement by Day 14 Maintained to Day 42
Description: Compare ≥2 category improvement on the WHO Ordinal Scale for Clinical Improvement from 0(uninfected) to 8(death) for subjects taking opaganib and those on placebo, lower scores indicate improvement. Success was defined as subject who reached improvement of at least two points on the WHO Ordinal Scale by Day 14, maintained by the end of study visit, and failure otherwise.
Time Frame: 14 days maintained up to 42 days
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 230 | 233
Participants
  Subject has improvement > or equal to 2 on the WHO Ordinal Scale Day 14 and up to to Day 42 | 145 | 138
  Subject has improvement of 1 or none on the WHO Ordinal Scale (Failure) Day 14 up to Day 42 | 85 | 95
  Failure due to not achieving improvement at Day 14: number analyzed (Participants) | 85 | 95
  Failure due to not achieving improvement at Day 14 | 64 | 69
  Failure due to death up to Day 14 (before any success): number analyzed (Participants) | 85 | 95
  Failure due to death up to Day 14 (before any success) | 18 | 21
  Failure due to missing status at Day 42 with prior success: number analyzed (Participants) | 85 | 95
  Failure due to missing status at Day 42 with prior success | 3 | 5
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.380, Cochran-Mantel-Haenszel — The threshold for statistical significance was p = 0.05, only if the primary endpoint was significant. This p-value is not adjusted for multiple comparisons because the primary endpoint was not met; Risk Difference (RD) = 3.91, 95% CI 2-sided [-4.78 to 12.60]

3. Secondary Outcome: Number of Subjects With Improvement to a Score of 3 or Less on the WHO Ordinal Scale for Clinical Improvement With a Scale Ranging From 8 Down to 0
Description: Compare scores of subjects taking opaganib and those on placebo, lower scores indicate improvement to determine time to recovery as defined by improvement to a score of 3 or less on the WHO Ordinal Scale for Clinical Improvement with a scale ranging from 0 (uninfected) to 8 (death)
Time Frame: 14 days maintained up to 42 days
Population: mITT population presenting subjects who experienced a recovery event by Day 14 maintained up to day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 230 | 233
Participants | 145 | 138
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.231, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.91 to 1.45]

4. Secondary Outcome: Number of Participants With Low Oxygen Flow Via Nasal Cannula
Description: To compare the time to low oxygen flow via nasal cannula e.g. from high oxygen flow via nasal cannula or CPAP, if high oxygen flow is not an available option between subjects taking opaganib and those on placebo.
Time Frame: 14 days maintained up to 42 days
Population: mITT. In this analysis, subjects who required low-flow supplemental oxygen at Day 1 (baseline) were considered success events, and the time to event of interest for these subjects was defined as 0.
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 230 | 233
Participants | 169 | 167
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.472, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio, log = 1.08, 95% CI 2-sided [0.87 to 1.33]

5. Secondary Outcome: Time to Discharge From Hospital Measured at 14 Days
Description: Time to subject discharge from hospital
Time Frame: 14 days
Population: mITT
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 230 | 233
Days | 13.50 [12.00 to 15.00] | 14.00 [NA to NA] — Not achieved
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.521, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.080, 95% CI 2-sided [0.846 to 1.378]

6. Secondary Outcome: Patients Requiring Intubation and Mechanical Ventilation by Day 42
Description: To compare the proportion of patients requiring intubation and mechanical ventilation between subjects taking opaganib and those on placebo.
Time Frame: 42 days
Population: Subjects requiring intubation by Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 230 | 233
Participants
  Subjects requiring intubation and mechanical ventilation by Day 42 (Failure) | 53 | 57
  Subjects not requiring intubation and mechanical ventilation by Day 42 (Success) | 177 | 176
  Type of failure: Intubation without death: number analyzed (Participants) | 53 | 57
  Type of failure: Intubation without death | 10 | 10
  Type of failure: Intubation with death: number analyzed (Participants) | 53 | 57
  Type of failure: Intubation with death | 33 | 33
  Type of failure: Death without intubation: number analyzed (Participants) | 53 | 57
  Type of failure: Death without intubation | 3 | 5
  Type of failure: Early termination/missing data (alive without intubation): number analyzed (Participants) | 53 | 57
  Type of failure: Early termination/missing data (alive without intubation) | 7 | 9
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.701, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = -1.51, 95% CI 2-sided [-9.19 to 6.18]

7. Secondary Outcome: Number of Patients With Two Consecutive Negative Swabs for SARS-CoV-2 at Day 14
Description: To compare the number of patients with two consecutive negative swabs for SARS-CoV-2 by PCR at Day 14 between subjects taking opaganib and those on placebo.
Time Frame: 14 days
Population: Only subjects who were positive for SARS-CoV-2 by PCR at the screening visit were analyzed
Measure: Number; unit: participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 218 | 219
participants
  Number of participants | 93 | 79
  Number of censored participants (observations) | 125 | 140
  Participants with no post baseline results available: number analyzed (Participants) | 125 | 140
  Participants with no post baseline results available | 13 | 8
  Participants with less than two results and discharged by Day 5: number analyzed (Participants) | 125 | 140
  Participants with less than two results and discharged by Day 5 | 7 | 7
  Participants with less than two results and not discharged by Day 5: number analyzed (Participants) | 125 | 140
  Participants with less than two results and not discharged by Day 5 | 21 | 24
  Participants with at least two results which are not two sequential negatives: number analyzed (Participants) | 125 | 140
  Participants with at least two results which are not two sequential negatives | 84 | 101
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority — The threshold for statistical significance was p = 0.05, only if the primary endpoint was significant. This p-value is not adjusted for multiple comparisons because the primary endpoint was not met; p = 0.043, Log Rank; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [0.99 to 1.82]

8. Secondary Outcome: Patients With Negative Swabs for SARS-CoV-2 at Day 14
Description: To compare the proportion of patients with two consecutive negative swabs for SARS-CoV-2 by PCR at Day 14 between subjects taking opaganib and those on placebo.
Time Frame: 14 days
Population: Only subjects who were positive for SARS-CoV-2 by PCR at the screening visit AND had at least two post baseline PCR tests were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 177 | 180
Participants
  Participants without two consecutive negative swabs for SARS-CoV-2 by PCR at Day 14 (Failure) | 93 | 79
  Participants with at least two consecutive negative swabs for SARS-CoV-2 by PCR at Day 14 (Success) | 84 | 101
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.118, Cochran-Mantel-Haenszel; Risk Difference (RD) = 8.30, 95% CI 2-sided [-2.05 to 18.65]

9. Secondary Outcome: Mortality Due to Any Cause
Description: To compare mortality 28 days post-baseline between subjects taking opaganib and those taking placebo
Time Frame: 28 days
Population: Mortality ("failure") was assessed by treatment Day 28 (including). Any early termination/ missing survival status at the end of study visit was also regarded as failure for the primary analysis of this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 230 | 233
Participants
  Yes (Failure) - Mortality due to any cause at Day 28 | 38 | 44
  No (Success) | 192 | 189

10. Secondary Outcome: Mortality Due to Any Cause
Description: To compare mortality 42 days post-baseline between subjects taking opaganib and those taking placebo
Time Frame: 42 days
Population: Mortality ("failure") was assessed by treatment Day 42 (including). Any early termination/ missing survival status at the end of study visit was also regarded as failure for the primary analysis of this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 230 | 233
Participants
  Yes (Failure) - Mortality due to any cause at Day 42 | 44 | 47
  No (Success) | 186 | 186

11. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: To compare the number of participants with treatment emergent adverse events (TEAEs) in patients with severe COVID-19 pneumonia between participants taking opaganib and participants taking placebo
Time Frame: From first dose until 4 weeks follow-up after the end of treatment
Population: TEAE=Treatment emergent adverse event. Treatment emergent events are events that started on or after the date of first dose
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 230 | 233
Participants | 155 | 147

12. Post Hoc Outcome: Supplemental Oxygen Requirement in the ≤60% FiO2 Sub-population
Description: Percentage of Subjects No Longer Requiring Supplemental Oxygen, for at Least 24 Hours by Day 14 in the ≤60% FiO2 FiO2 Sub-populations
Time Frame: Day 14
Population: A post hoc analysis set comprised two sub-populations, namely, "lower FiO2" (FiO2 at baseline ≤ the median of 60%) and "higher FiO2" (FiO2 at baseline > the median of 60%) was added after the final version of the SAP was signed.
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 117 | 134
Participants
  Subjects no longer requiring oxygen for at least 24 hours by Day 14 | 90 | 85
  Subjects requiring oxygen (including death, lost to follow-up or need of oxygen) | 27 | 49
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.033, Cochran-Mantel-Haenszel — unadjusted p-value; Risk Difference (RD) = 12.28, 95% CI 2-sided [1.06 to 23.50]

13. Post Hoc Outcome: Supplemental Oxygen Requirement in the > 60% FiO2 Sub-population
Description: Percentage of Subjects No Longer Requiring Supplemental Oxygen, for at Least 24 Hours by Day 14 in the > 60% FiO2 FiO2 Sub-populations
Time Frame: Day 14
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 105 | 88
Participants
  Subjects no longer requiring oxygen for at least 24 hours by Day 14 | 43 | 41
  Subjects requiring oxygen (including death, lost to follow-up or need of oxygen) | 62 | 47
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.500, Cochran-Mantel-Haenszel; Risk Difference (RD) = -4.75, 95% CI 2-sided [-18.67 to 9.17]

14. Post Hoc Outcome: Subjects With ≥ 2 Category Improvement on the WHO Ordinal Scale for Clinical Improvement by Day 14 Maintained to Day 42 in the FiO2 ≤ 60% Population
Description: Post hoc analysis in the FiO2 ≤ 60% population. Compare ≥2 category improvement on the WHO Ordinal Scale for subjects taking opaganib and those on placebo, lower scores indicate improvement. Success was defined as subject who reached improvement of at least two points on the WHO Ordinal Scale by Day 14, maintained by the end of study visit day 42, and failure otherwise. WHO Ordinal Scale for Clinical Improvement is a scale from 0 (uninfected) to 8 (death) with higher scale poorer clinical status
Time Frame: 14 days maintained up to 42 days or classified as a failure
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 117 | 134
Participants
  Subject has improvement of 2 or more on the WHO Ordinal Scale (Success) Day 14 maintained to day 42 | 93 | 88
  Subject has improvement of 1 or does not show improvement on the WHO Ordinal Scale (Failure) Day 14 | 24 | 46
  Failure due to not achieving improvement at Day 14: number analyzed (Participants) | 24 | 46
  Failure due to not achieving improvement at Day 14 | 21 | 29
  Failure due to death up to Day 14 (before any success): number analyzed (Participants) | 24 | 46
  Failure due to death up to Day 14 (before any success) | 3 | 13
  Failure due to missing status at Day 42 with prior success at Day 14: number analyzed (Participants) | 24 | 46
  Failure due to missing status at Day 42 with prior success at Day 14 | 0 | 4
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.023, Cochran-Mantel-Haenszel; Risk Difference (RD) = 12.75, 95% CI 2-sided [1.90 to 23.60]

15. Post Hoc Outcome: Subjects With ≥ 2 Category Improvement on the WHO Ordinal Scale for Clinical Improvement by Day 14 up to Day 42 in the FiO2 > 60% Population
Description: Post hoc analysis in the FiO2 > 60% population. Compare ≥2 category improvement on the WHO Clinical Ordinal Scale for subjects taking opaganib and those on placebo, lower scores indicate improvement. Success was defined as subject who reached improvement of at least two points on the WHO Ordinal Scale by Day 14, maintained by the end of study visit day 42 and failure otherwise.WHO Scale 0 to 8 with 8 death and higher number worse clinical state
Time Frame: 14 days maintained up to 42 days or classifed as failure
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 105 | 88
Participants
  Subject has improvement of 2 or more on the WHO Ordinal Scale (Success) Day 14 maintained to Day 42 | 46 | 43
  Subject has improvement of 1 or no improvement shown on the WHO Ordinal Scale (Failure) at Day 14 | 59 | 45
  Failure due to not achieving improvement at Day 14: number analyzed (Participants) | 59 | 45
  Failure due to not achieving improvement at Day 14 | 41 | 37
  Failure due to death up to Day 14 (before any success): number analyzed (Participants) | 59 | 45
  Failure due to death up to Day 14 (before any success) | 15 | 7
  Failure due to missing status at Day 42 with prior success: number analyzed (Participants) | 59 | 45
  Failure due to missing status at Day 42 with prior success | 3 | 1
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.561, Cochran-Mantel-Haenszel; Risk Difference (RD) = -4.12, 95% CI 2-sided [-18.07 to 9.82]

16. Post Hoc Outcome: Number of Subjects With Improvement to a Score of 3 or Less on the WHO Ordinal Scale for Clinical Improvement in the FiO2 ≤60% Population
Description: Compare scores of subjects taking opaganib and those on placebo, lower scores indicate improvement.
  WHO Ordinal Scale for Clinical Improvement with a scale ranging from 8 down to 0 with a higher score indicating a poorer clinical status
Time Frame: 14 days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 117 | 134
Participants | 93 | 88
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.01, Log Rank; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [1.07 to 1.93]

17. Post Hoc Outcome: Number of Subjects With Improvement to a Score of 3 or Less on the WHO Ordinal Scale for Clinical Improvement in the FiO2 > 60% Population
Description: Compare scores of subjects taking opaganib and those on placebo, lower scores indicate improvement.
  World Health Organization Ordinal Scale for Clinical Improvement with a scale ranging from 8 down to 0 with a higher score indicating poorer clincal status
Time Frame: 14 days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 105 | 88
Participants | 46 | 43
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.545, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.58 to 1.34]

18. Post Hoc Outcome: Number of Subjects Discharged From Hospital in the FiO2 ≤60% Population
Description: Subjects discharged from the hospital in the FiO2 ≤60% population at 14 days
Time Frame: 14 days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 117 | 134
Participants | 81 | 85
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.100, Log Rank; Hazard Ratio (HR) = 1.276, 95% CI 2-sided [0.940 to 1.732]

19. Post Hoc Outcome: Number of Subjects Discharged From Hospital in the FiO2 > 60% Population
Description: Number of subjects discharged from the hospital in the FiO2 > 60% population
Time Frame: 14 days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 105 | 88
Participants | 41 | 40

20. Post Hoc Outcome: Requiring Intubation and Mechanical Ventilation by Day 42 in the FiO2 ≤60% Population
Description: To compare the proportion of patients in the FiO2 ≤60% sub-population requiring intubation and mechanical ventilation between subjects taking opaganib and those on placebo.
Time Frame: 42 days
Population: Subjects requiring intubation by Day 42 in the FiO2 ≤60% sub-population
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 117 | 134
Participants
  Subjects requiring intubation and mechanical ventilation by Day 42 (Failure) | 8 | 24
  Subjects not requiring intubation and mechanical ventilation by Day 42 (Success) | 109 | 110
  Type of failure: Intubation without death: number analyzed (Participants) | 8 | 24
  Type of failure: Intubation without death | 2 | 3
  Type of failure: Intubation with death: number analyzed (Participants) | 8 | 24
  Type of failure: Intubation with death | 5 | 15
  Type of failure: Death without intubation: number analyzed (Participants) | 8 | 24
  Type of failure: Death without intubation | 0 | 1
  Type of failure: Early termination/missing data (alive without intubation): number analyzed (Participants) | 8 | 24
  Type of failure: Early termination/missing data (alive without intubation) | 1 | 5
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.012, Cochran-Mantel-Haenszel; Risk Difference (RD) = -10.50, 95% CI 2-sided [-18.44 to -2.57]

21. Post Hoc Outcome: Requiring Intubation and Mechanical Ventilation by Day 42 in the FiO2 > 60% Population
Description: To compare the proportion of patients in the FiO2 > 60% sub-population requiring intubation and mechanical ventilation between subjects taking opaganib and those on placebo.
Time Frame: 42 days
Population: Subjects requiring intubation by Day 42 in the FiO2 ≤60% sub-population
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 105 | 88
Participants
  Subjects requiring intubation and mechanical ventilation by Day 42 (Failure) | 43 | 30
  Subjects not requiring intubation and mechanical ventilation by Day 42 (Success) | 62 | 58
  Type of failure: Intubation without death: number analyzed (Participants) | 43 | 30
  Type of failure: Intubation without death | 7 | 6
  Type of failure: Intubation with death: number analyzed (Participants) | 43 | 30
  Type of failure: Intubation with death | 28 | 16
  Type of failure: Death without intubation: number analyzed (Participants) | 43 | 30
  Type of failure: Death without intubation | 3 | 4
  Type of failure: Early termination/missing data (alive without intubation): number analyzed (Participants) | 43 | 30
  Type of failure: Early termination/missing data (alive without intubation) | 5 | 4
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.304, Cochran-Mantel-Haenszel; Risk Difference (RD) = 7.20, 95% CI 2-sided [-6.46 to 20.86]

22. Post Hoc Outcome: Mortality Due to Any Cause in the FiO2 ≤60% Population
Description: To compare mortality 28 and 42 days post-baseline between subjects taking opaganib and those taking placebo in the in the FiO2 ≤60% population
Time Frame: 28 and 42 days
Population: Mortality ("failure") was assessed by treatment Day 28 (including) and Day 42. Any early termination/ missing survival status at the end of study visit was also regarded as failure for the primary analysis of this endpoint.
  For the FiO2 ≤60% Sub-population
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 117 | 134
Participants
  Mortality due to any cause at Day 28 in the FiO2 ≤60% population: Yes (Failure) - Mortality due to any cause | 7 | 21
  Mortality due to any cause at Day 28 in the FiO2 ≤60% population: No (Success) | 110 | 113
  Mortality due to any cause at Day 42 in the FiO2 ≤60% population: Yes (Failure) - Mortality due to any cause | 7 | 21
  Mortality due to any cause at Day 42 in the FiO2 ≤60% population: No (Success) | 110 | 113
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.019, Cochran-Mantel-Haenszel; Risk Difference (RD) = -9.22, 95% CI 2-sided [-16.63 to -1.80]

23. Post Hoc Outcome: Mortality Due to Any Cause in the FiO2 > 60% Population
Description: To compare mortality 28 and 42 days post-baseline between subjects taking opaganib and those taking placebo in the in the FiO2 > 60% population
Time Frame: 28 and 42 days
Population: Mortality ("failure") was assessed by treatment Day 28 (including) and Day 42. Any early termination/ missing survival status at the end of study visit was also regarded as failure for the primary analysis of this endpoint.
  For the FiO2 > 60% Sub-population
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 105 | 88
Participants
  Mortality due to any cause at Day 28 in the FiO2 > 60% population: Yes (Failure) | 30 | 21
  Mortality due to any cause at Day 28 in the FiO2 > 60% population: No (Success) | 75 | 67
  Mortality due to any cause at Day 42 in the FiO2 > 60% population: Yes (Failure) | 36 | 24
  Mortality due to any cause at Day 42 in the FiO2 > 60% population: No (Success) | 69 | 64
Statistical Analysis 1: Comparison: Opaganib vs Placebo; Test type: Superiority; p = 0.273, Cochran-Mantel-Haenszel; Risk Difference (RD) = 7.37, 95% CI 2-sided [-5.66 to 20.39]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first study drug dose (Day 1) until 4 weeks follow-up after the end of treatment, up to 42 days
Description: TEAE=Treatment emergent adverse event. Treatment emergent events are adverse events that started on or after the date of first dose.
Groups:
- Opaganib: Standard of care + opaganib, 2 x 250 mg oral capsules (500 mg), every 12 hours, for 14 days (Day 1 to Day 14).
- Placebo: Standard of care + matching placebo, 2 x 250 mg oral capsules (500 mg), every 12 hours, for 14 days (Day 1 to Day 14).
Arm/Group | Opaganib | Placebo
All-Cause Mortality (participants affected / at risk) | 44/230 | 47/233
Serious Adverse Events (participants affected / at risk) | 52/230 | 52/233
Other Adverse Events (participants affected / at risk) | 155/230 | 147/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opaganib (N=230) | Placebo (N=233)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 13 (13)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cerebral thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Femoral artery embolism (Vascular disorders) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 10 (11) | 6 (7)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 16 (16)
Sepsis (Infections and infestations) | 2 (2) | 7 (7)
Septic shock (Infections and infestations) | 5 (5) | 6 (6)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opaganib (N=230) | Placebo (N=233)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (4) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Administration site phlebitis (General disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 12 (12) | 14 (14)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (8) | 3 (3)
Anxiety (Psychiatric disorders) | 8 (8) | 3 (3)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 4 (4)
Asthenia (General disorders) | 1 (1) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 5 (8) | 3 (3)
Axillary vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 3 (3)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood lactic acid increased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood pressure diastolic decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 4 (5)
Blood sodium increased (Investigations) | 1 (1) | 0 (0)
Blue toe syndrome (Vascular disorders) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 2 (2) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cerebral atrophy (Nervous system disorders) | 1 (1) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 22 (23) | 24 (24)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 3 (3) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 6 (6)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 7 (8) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 3 (3) | 4 (4)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Enterococcus test positive (Investigations) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 0 (0) | 2 (2)
Eye irritation (Eye disorders) | 1 (1) | 1 (1)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haemochromatosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 8 (8) | 4 (4)
Hepatic enzyme increased (Investigations) | 2 (2) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis B core antibody positive (Investigations) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 2 (2) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 9 (9) | 8 (11)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 4 (5) | 6 (6)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 7 (8) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Inflammatory marker increased (Investigations) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 17 (18) | 9 (9)
Interleukin level increased (Investigations) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella test positive (Investigations) | 0 (0) | 2 (2)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Mechanical ventilation (Surgical and medical procedures) | 1 (1) | 1 (1)
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Myopia (Eye disorders) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (13) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 6 (6) | 5 (5)
Oral candidiasis (Infections and infestations) | 2 (2) | 8 (8)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 5 (5)
Pain (General disorders) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Persistent depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 3 (3) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (6) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia necrotising (Infections and infestations) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Post intensive care syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 2 (2)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Pupils unequal (Eye disorders) | 0 (0) | 1 (1)
Purulent discharge (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 7 (8) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (7)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Scrotal dermatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Serratia infection (Infections and infestations) | 0 (0) | 1 (1)
Serum ferritin increased (Investigations) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 4 (4)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sputum purulent (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 3 (3) | 0 (0)
Steroid diabetes (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 4 (4) | 11 (15)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 4 (5)
Thrombophlebitis (Vascular disorders) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tongue discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 4 (4)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 6 (6)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT04467840/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT04467840/SAP_001.pdf